CLINICAL TRIAL: NCT04347018
Title: Alignment and Discomfort Using Non-Sliding Lingual Orthodontic Technique (BRIUS) and Conventional Bracket Systems: A Single-Center Randomized Clinical Trial
Brief Title: BRIUS Vs FFA Efficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Mohammed H Al-Zainal, Orthodontic Resident, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRvFFA
Record Dates: First submitted 2020-04-12; First posted 2020-04-15 (Actual); Results first posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-09

CONDITIONS: Dental Malocclusion; Angle Class II; Angle Class I; Crowding, Tooth
MeSH Terms: conditions — Malocclusion; Malocclusion, Angle Class II; Malocclusion, Angle Class I

STUDY DESIGN:
Intervention Model Description: 2 groups will receive treatment and be observed over the course of the alignment phase of their orthodontic treatment. Regular photographic records will be taken during appointments and the data will be analysed after the 18 week period is completed for all patients involved in the study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BRIUS (Experimental): BRIUS orthodontic appliance (wire) will be used to treat the patients. BRIUS appliance will be engaged to regular orthodontic brackets intra-orally to initiate orthodontic treatment at the University at Buffalo Orthodontic Clinic.
  Interventions: Device: BRIUS
- Preadjusted edgewise full fixed appliance (Active Comparator): regular full fixed orthodontic appliance (FFA) appliances will be used to treat patients. These are regular orthodontic brackets with standard orthodontic wires used to treat patients at the University at Buffalo Department of Orthodontics
  Interventions: Device: BRIUS

INTERVENTIONS:
Device: BRIUS — This is a device that is designed based on movements planned virtually on a computer program. Then all the planned movements are embedded into the wire causing the wire to have the necessary bends to move every tooth into its pre-planned final position. This causes the pre-activated wire to consistently express a low force over a long period of time onto all the teeth. This allows the teeth to move into the final position and treatment progresses towards completion

SUMMARY:
The purpose of this study is to compare the Full Fixed Preadjusted appliances (regular braces) when to the BRIUS system.

DETAILED DESCRIPTION:
This is a randomized controlled trial which aims to identify the effectiveness of alignment in the BRIUS group when compared to the full fixed appliance group.

The secondary aim of the study is to identify any difference in discomfort experienced by the patients when undergoing treatment using the two appliances

The investigators also aim to quantify the extent of tooth movement that is achieved through each appliance within a given time frame

ELIGIBILITY:
Inclusion Criteria:

* 10 to 18 years old
* Angle Class I and Cl II (up to half cusp) molar and canine relationship.
* Fully erupted permanent dentition (excluding third molars).
* Crowding of 7 mm or less.
* Must be able to maintain good oral hygiene assessed by the orthodontist during their visits.

Exclusion Criteria:

* Previous history of orthodontic treatment or orthognathic surgery
* Subjects who require extractions or orthognathic surgery
* Multiple missed appointments
* Deteriorating oral hygiene and craniofacial syndromes or disorders
* Severe gag reflex resulting from the use of intra-oral scanners

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed h alzainal, BDS, Principal Investigator — Orthodontic resident
Locations (1):
- Department of Orthodontics, School of Dental Medicine, SUNY at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] S.M.R. Peikar, J.S. Wratten Jr, Teeth repositioning systems and methods, Google Patents, 2019.
- [Background] Ioshida M, Munoz BA, Rios H, Cevidanes L, Aristizabal JF, Rey D, Kim-Berman H, Yatabe M, Benavides E, Alvarez MA, Volk S, Ruellas AC. Accuracy and reliability of mandibular digital model registration with use of the mucogingival junction as the reference. Oral Surg Oral Med Oral Pathol Oral Radiol. 2019 Apr;127(4):351-360. doi: 10.1016/j.oooo.2018.10.003. Epub 2018 Oct 16. PMID 30472195
- [Background] Grauer D, Proffit WR. Accuracy in tooth positioning with a fully customized lingual orthodontic appliance. Am J Orthod Dentofacial Orthop. 2011 Sep;140(3):433-43. doi: 10.1016/j.ajodo.2011.01.020. PMID 21889089
- [Result] Scott P, DiBiase AT, Sherriff M, Cobourne MT. Alignment efficiency of Damon3 self-ligating and conventional orthodontic bracket systems: a randomized clinical trial. Am J Orthod Dentofacial Orthop. 2008 Oct;134(4):470.e1-8. doi: 10.1016/j.ajodo.2008.04.018. PMID 18929262
- [Result] Wu AK, McGrath C, Wong RW, Wiechmann D, Rabie AB. A comparison of pain experienced by patients treated with labial and lingual orthodontic appliances. Eur J Orthod. 2010 Aug;32(4):403-7. doi: 10.1093/ejo/cjp117. Epub 2009 Dec 16. PMID 20018798
- [Result] Wu A, McGrath C, Wong RW, Wiechmann D, Rabie AB. Comparison of oral impacts experienced by patients treated with labial or customized lingual fixed orthodontic appliances. Am J Orthod Dentofacial Orthop. 2011 Jun;139(6):784-90. doi: 10.1016/j.ajodo.2009.07.027. PMID 21640885
- [Result] Talaat S, Kaboudan A, Bourauel C, Ragy N, Kula K, Ghoneima A. Validity and reliability of three-dimensional palatal superimposition of digital dental models. Eur J Orthod. 2017 Aug 1;39(4):365-370. doi: 10.1093/ejo/cjx008. PMID 28339627

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BRIUS | Preadjusted Edgewise Full Fixed Appliance
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BRIUS | Preadjusted Edgewise Full Fixed Appliance | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 13
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 3 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Overall 3D Movement
Description: absoluate measurement of extent of movement of teeth
Time Frame: 18 weeks
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | BRIUS | Preadjusted Edgewise Full Fixed Appliance
Number analyzed (Participants) | 7 | 6
mm | 1.46 [0.16 to 2] | 1.41 [0.15 to 2.56]

2. Primary Outcome: Little's Irregularity Index
Description: Little's irregularity index. The index measures the alignment discrepancy in the five contact points of the lower anterior region in millimeteres. The minimum score is zero and the maximum is 10 or above. The greater the score the worse the outcome
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | BRIUS | Preadjusted Edgewise Full Fixed Appliance
Number analyzed (Participants) | 7 | 6
Millimeter | 5.38 (3.04) | 5.04 (1.61)

3. Primary Outcome: Discomfort
Description: Online survey will evaluate discomfort arising from the orthodontic brackets between patients in the two groups. A visual analog scale from 0-10 millimeter will be applied. The greater the score the worse the discomfort level.
Time Frame: 18 weeks
Measure: Mean (Inter-Quartile Range); unit: units on a scale - millimeter
Arm/Group | BRIUS | Preadjusted Edgewise Full Fixed Appliance
Number analyzed (Participants) | 7 | 6
units on a scale - millimeter | 1.57 [0 to 7] | 38.67 [21 to 59]

ADVERSE EVENTS:
Time Frame: 18 weeks
Description: None of the participants had any risk factors that could cause serious adverse events or mortality
Arm/Group | BRIUS | Preadjusted Edgewise Full Fixed Appliance
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT04347018/Prot_SAP_000.pdf